CLINICAL TRIAL: NCT02327715
Title: Emtricitabine for Prevention of Vertical Transmission of HBV in Chinese Pregnant HBsAg Positive Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asian-Pacific Alliance of Liver Disease, Beijing (Other)
Collaborators: Beijing Ditan Hospital (Other); Hebei Medical University Pharmaceutical Factory (Industry); National Health and Family Planning Commission, P.R.China (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FTC-02-prevention
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Hepatitis B, Chronic; Pregnancy
Keywords: Hepatitis B virus; Emtricitabine; Pregnancy; Vertical transmission
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chinese naive pregnant HBsAg positive patients (Experimental): single group patients were enrolled to receive emtricitabine(200mg one time per day) till 24 weeks after dilivery,patients and followed up for 24 weeks.
  Interventions: Drug: Emtricitabine

INTERVENTIONS:
Drug: Emtricitabine — emtricitabine were given to each patients from week 28 pregnancy to 24 weeks after delivery
  Other Names: Brand name：Huierding

SUMMARY:
This study evaluates generic emtricitabine(FTC) efficacy and safety in Chinese naive pregnant HBsAg positive patients in prevention of HBV vertical transmission. Single group patients were enrolled to receive emtricitabine till 24 weeks after delivery.

DETAILED DESCRIPTION:
Single group patients were enrolled to receive emtricitabine till 24 weeks after delivery, which include HBeAg positive patients. Patients and their newborns were followed till 48 weeks after delivery to evaluate the efficacy of prevention of vertical transmission.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive for more than 6 months
* HBeAg positive patients: HBV DNA ≥ 5log10 copies/ml
* HBeAg postive patients: ALT≥2×ULN;or liver biopsy G≥2;or liver biopsy S ≥2;or liver biopsy Knodell HAI ≥ 4
* HBeAg negative patients: HBV DNA ≥ 4log10 copies/ml
* HBeAg postive patients: ALT≥2×ULN;or liver biopsy G≥2;or liver biopsy S ≥2;or liver biopsy Knodell HAI ≥ 4
* Nucleoside/nucleotide naive paitents
* Diagnosed as ≥ 28 weeks pregnancy

Exclusion Criteria:

* Diagnosed HCC with AFP and ultrasound, CT or MRI
* Creatine >130μmol/L or Ccr < 70mL/min
* Hemoglobin <100g/L
* Coinfected with HAV,HEV,HCV,HDV or HIV
* ANA > 1:100
* Uncontrolled cardiovascluar diseases, kidney diseases,lung diseases, neurological diseases, digestive diseases,metabolic disorders, immune-compromised diseases or cancer
* Drug abuse or alcohal addiction
* Previous history of taking agents of lamivudine, adefovir, tenofovir entecavir or telbivudine
* Long-term use of immunosuppressor or immunomodulator 6 months before enrollment to this trial
* Underwent liver transplantation or liver transplantation in schedule
* Allergic to nucleoside or nucleotide analogues
* family history of genetic defects disease
* Abnormal results in fatal defects screening
* HBsAg positive sperm provider pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
HBsAg positive rate in newborns | week48 after delivery
  HBsAg positive rate in newborns

SECONDARY OUTCOMES:
birth defect in newborns | 0 weeks, week24 and week48 after delivery
  birth defect in newborns
virological response rate | week 24 after delivery
  HBV DNA < 500 copies/ml
HBV DNA decrease level | week 24 after delivery
  HBV DNA decrease compared with baseline（log10 copies/ml）
biochemical response | week 24 after delivery
  ALT normalization
HBeAg loss | week 24 after delivery
  HBeAg loss in HBeAg positive patients
HBeAg seroconversion | week 24 after delivery
  HBeAg seroconversion in HBeAg positive group
HBV genetic resistance to emtricitabine | week 24 after delivery
  HBV genetic resistance to emtricitabine
adverse event | week 24 after delivery
  type and rate of adverse events;type and rate of severe adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cheng, M.D., Principal Investigator — Asian Pacific Alliance of Liver Diseases, Beijing

REFERENCES:
- [Background] Gish RG, Leung NW, Wright TL, Trinh H, Lang W, Kessler HA, Fang L, Wang LH, Delehanty J, Rigney A, Mondou E, Snow A, Rousseau F. Dose range study of pharmacokinetics, safety, and preliminary antiviral activity of emtricitabine in adults with hepatitis B virus infection. Antimicrob Agents Chemother. 2002 Jun;46(6):1734-40. doi: 10.1128/AAC.46.6.1734-1740.2002. PMID 12019083
- [Background] Lim SG, Ng TM, Kung N, Krastev Z, Volfova M, Husa P, Lee SS, Chan S, Shiffman ML, Washington MK, Rigney A, Anderson J, Mondou E, Snow A, Sorbel J, Guan R, Rousseau F; Emtricitabine FTCB-301 Study Group. A double-blind placebo-controlled study of emtricitabine in chronic hepatitis B. Arch Intern Med. 2006 Jan 9;166(1):49-56. doi: 10.1001/archinte.166.1.49. PMID 16401810